CLINICAL TRIAL: NCT01330030
Title: Selegiline Patch for Treatment of Nicotine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joel D Killen, Principle Investigator, Stanford University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SU-07232007-459; R01DA017457 (NIH); NCT00218647 (obsolete NCT alias)
Record Dates: First submitted 2010-11-08; First posted 2011-04-06 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-05

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Selegiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug Selegiline (Experimental): 6 mg selegiline patch (transdermal) worn for 24 hours for 8 weeks
  Interventions: Drug: Selegiline
- Matching placebo (Placebo Comparator): matching placebo worn 24 hours for 8 weeks
  Interventions: Other: matching placebo

INTERVENTIONS:
Drug: Selegiline — 6mg/24 hrs for 8 weeks
  Other Names: EMSAM
  Arms: Drug Selegiline
Other: matching placebo — placebo/24hrs for 8 weeks
  Other Names: Placebo
  Arms: Matching placebo

SUMMARY:
Relapse to smoking is a common problem affecting smokers who seek treatment. The purpose of this study is examine whether selegiline, given in the form of a skin patch, is effective in stopping smoking.

DETAILED DESCRIPTION:
Most smokers relapse following smoking cessation treatment. More effective smoking cessation therapies are needed to prevent the high rates of relapse. Selegiline is a selective inhibitor of monoamine oxidase B (MAO B) and has been used clinically in combination with levodopa to treat Parkinson's disease. Selegiline permits the stabilization of dopamine (DA) levels in the brain by preventing the rapid degradation of DA by means of MAO B and is used as an adjunct to levodopa therapy causing a dose-sparing effect and enhancing dopaminergic transmission. Selegiline's effect on MAO B and the resulting effect on brain DA has interesting implications for the treatment of nicotine dependence because brain DA systems may play a key role in the mediation of reward learning behavior. Previous research suggests that the brains of living smokers show a 40% decrease in the level of MAO B relative to nonsmokers or former smokers. The purpose of this study is examine whether selegiline, administered in the form of a skin patch, is effective for smoking cessation.

Participants will be randomly assigned to one of two treatments: 1) transdermal selegiline patch (STS) or 2) placebo. Treatment with STS or placebo will be given for a period of 8 weeks. Participants will be stratified by gender to evaluate the role that gender plays in moderating smoking cessation treatment. Study visits will take place once each week for 30 to 45 minutes, and will include adverse events monitoring, biochemical verification of smoking status, and a physical exam. Follow-up visits will occur at Weeks 24 and 52 to determine response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Smokes greater than 20 cigarettes per day

Exclusion Criteria:

* History of Parkinson's disease, high blood pressure, or severe liver or kidney disease
* Current substance abuse
* Mental illness
* Skin conditions that could interfere with patch use
* Using antidepressant medications (e.g., levodopa/carbidopa, methyldopa, or any MAO inhibitor)
* Pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2005-07; Primary Completion 2008-08 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel D Killen, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Killen JD, Fortmann SP, Murphy GM Jr, Hayward C, Fong D, Lowenthal K, Bryson SW, Killen DT, Schatzberg AF. Failure to improve cigarette smoking abstinence with transdermal selegiline + cognitive behavior therapy. Addiction. 2010 Sep;105(9):1660-8. doi: 10.1111/j.1360-0443.2010.03020.x. PMID 20707784
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The original target enrollment was 230. Over recruitment led to a study sample size =243
Period: Overall Study
Arm/Group | Drug Selegiline | Matching Placebo
Started | 121 | 122
Completed | 105 (number assessed at week 52 follow-up) | 105 (number assessed at week 52 follow-up)
Not Completed | 16 | 17
Not completed — Lost to Follow-up | 16 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug Selegiline | Matching Placebo | Total
Number analyzed (Participants) | 121 | 122 | 243
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 121 | 122 | 243
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 74
  Male | 84 | 85 | 169
Region of Enrollment [Number; unit: participants]
  United States | 121 | 122 | 243

OUTCOME MEASURES:

1. Primary Outcome: Expired-air Carbon Monoxide Confirmed Smoking Abstinence
Description: expired-air carbon monoxide confirmed smoking abstinence at 52 weeks
Time Frame: 52 weeks
Population: intention to treat
Measure: Number; unit: participants not smoking
Arm/Group | Drug Selegiline | Matching Placebo
Number analyzed (Participants) | 121 | 122
participants not smoking | 24 | 25

ADVERSE EVENTS:
Arm/Group | Drug Selegiline | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 0/121 | 0/122
Other Adverse Events (participants affected / at risk) | 110/121 | 108/122
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug Selegiline (N=121) | Matching Placebo (N=122)
Insomnia (Psychiatric disorders) | 57 (57) | 53 (53)
Headache (General disorders) | 41 (41) | 43 (43)
skin rash (Skin and subcutaneous tissue disorders) | 30 (30) | 27 (27)
racing thoughts (Psychiatric disorders) | 25 (25) | 28 (28)
Lightheaded (General disorders) | 20 (20) | 20 (20)
Vivid dreams (Psychiatric disorders) | 13 (13) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes